CLINICAL TRIAL: NCT00063232
Title: Treatment of Nonalcoholic Steatohepatitis With Metformin
Brief Title: Treating Nonalcoholic Steatohepatitis (NASH) With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jay Hoofnagle, M.D./National Institute of Diabetes and Digestive and Kidney Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 030233; 03-DK-0233
Record Dates: First submitted 2003-06-23; First posted 2003-06-24 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis
Keywords: Insulin; Obesity; Fatty Liver; Diabetes; Cirrhosis; Metformin; Insulin Resistance; Nonalcoholic Steatohepatitis; Hepatitis; NASH
MeSH Terms: conditions — Hepatitis; Insulin Resistance; Obesity; Fatty Liver; Diabetes Mellitus; Fibrosis; Non-alcoholic Fatty Liver Disease | interventions — Metformin

INTERVENTIONS:
Drug: Metformin — After complete medical evaluation and liver biopsy, patients who qualified for therapy were started on metformin in an initial dose of 500 mg once daily. After 2 weeks, the dose was increased to 500 mg twice daily and after 4 weeks to the full dose of 1000 mg twice daily. Subsequent dose reductions were carried out based on tolerance, with particular attention to gastrointestinal upset and abdominal bloating. Patients were seen in the out-patient clinic, had a brief medical history and examination and routine blood tests at 2 and 4 weeks after enrolment and every 4 weeks thereafter. The oral and intravenous glucose tolerance tests were repeated after 40 and 44 weeks respectively and liver biopsy and imaging tests at 48 weeks. Metformin was discontinued after 48 weeks in patients without diabetes on the pre-treatment evaluation.

SUMMARY:
Nonalcoholic Steatohepatitis (NASH) is associated with progressive liver disease, fibrosis, and cirrhosis. Although the cause of NASH is unknown, it is often associated with obesity, type 2 diabetes, and insulin resistance. At present, there are no approved treatments for NASH patients, but an experimental approach has focused on improving their insulin sensitivity. Metformin is one of the most commonly used medications for the treatment of diabetes.

The purpose of this study is to determine whether the medical problems of NASH patients, specifically liver damage, improves when their insulin sensitivity is enhanced with metformin.

The study will last 3 to 5 years and will enroll up to 30 patients. Participants will undergo a complete medical examination, a series of lab tests, and a liver biopsy. They will then start taking a single 500-mg tablet of metformin once a day for 2 weeks, then the same dosage twice a day for 2 more weeks, if they tolerate the first dosage. The dosage will increase to 1,000 mg twice a day for the remaining 44 weeks of the study. After 1 year, participants will undergo a repeat medical examination and liver biopsy.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) represents a spectrum of diseases ranging from simple fatty liver (steatosis) to steatosis with inflammation and necrosis to cirrhosis, that occurs in persons who drink little or no alcohol. Nonalcoholic steatohepatitis (NASH) represents the more severe end of this spectrum and is associated with progressive liver disease, fibrosis and cirrhosis. The etiology of NASH is unclear, but it is often associated with obesity, type 2 diabetes, hyperlipidemia and insulin resistance. We have recently conducted a study of a 48-week course of pioglitazone in 21 non-diabetic patients with NASH. Serum aminotransferase levels and liver histology improved in most patients and the improvements correlated with changes in insulin sensitivity. These results are promising, but pioglitazone is associated with significant weight gain, is quite expensive, and its long-term safety is yet to be proven. In contrast, metformin is inexpensive, extremely well tolerated, and of proven long-term safety in patients with diabetes and pre-diabetes.

In this study, we propose to treat 20 non-diabetic patients with NASH with metformin for 48-weeks. After an initial evaluation for insulin sensitivity, fat distribution and liver biopsy, patients will receive gradually increasing doses of metformin orally to a maximum of 2000 mg daily. Patients will be monitored at regular intervals for symptoms of liver disease, side effects of metformin and serum biochemical and metabolic indices. At the end of 48-weeks, patients will have a repeat medical evaluation and liver biopsy. Pre and post treatment liver histology, fat distribution and insulin sensitivity will be compared. The primary end point of successful therapy will be improvement in hepatic histology as determined by reduction of at least three points in NASH activity score. Secondary end points will be improvement in insulin sensitivity, body fat distribution, and liver biochemistry.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age at entry at least 18 years.
  2. Serum alanine (ALT) or aspartate (AST) aminotransferase activities that are above the upper limits of normal.
  3. Evidence of steatohepatitis on liver biopsy done within the previous 12 months with a NASH activity score of at least 4 (of a total possible score of 16) including a score of at least 1 each for steatosis, hepatocellular injury and parenchymal inflammation. Histological criteria of steatohepatitis include: (1) macrovesicular steatosis, (2) acinar zone 3 hepatocellular injury (ballooning degeneration), (3) parenchymal and (4) portal inflammation. Additionally helpful, but not required, features include the presence of (5) Mallory's hyaline and (6) pericellular and/or sinusoidal fibrosis that predominantly involves zone 3.
  4. Written informed consent.

EXCLUSION CRITERIA:

1. Evidence of another form of liver disease.

   1. Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
   2. Hepatitis C as defined by presence of hepatitis C virus (HCV) RNA in serum.
   3. Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
   4. Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
   5. Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
   6. Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
   7. Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
   8. Drug-induced liver disease as defined on the basis of typical exposure and history.
   9. Bile duct obstruction as shown by imaging studies.
2. History of excess alcohol ingestion, averaging more than 30 gm/day (3 drinks per day) in the previous 10 years, or history of alcohol intake averaging greater than 10 gm/day (1drink per day: 7 drinks per week) in the previous one year.
3. Contraindications to liver biopsy: platelet counts less than 75,000/mm(3) or prothrombin time greater than 16 seconds.
4. Decompensated liver disease, Child-Pugh score greater than or equal to 7 points.
5. History of gastrointestinal bypass surgery or ingestion of drugs known to produce hepatic steatosis including corticosteroids, high-dose estrogens, methotrexate, tetracycline or amiodarone in the previous 6 months.
6. Presence of diabetes mellitus as defined by: fasting plasma glucose of greater than or equal to 126 mg/dl on two separate occasion, or diabetic symptoms with a random plasma glucose of greater than or equal to 200 mg/dl (34).
7. Use of anti-diabetic drugs, including insulin, biguanides, sulfonylureas, or thiazolidinediones in the previous 6 months.
8. Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease with hypoxia, renal failure, organ transplantation, serious psychiatric disease, malignancy that, in the opinion of the investigator would preclude treatment with metformin and adequate follow up.
9. Positive test for anti-HIV.
10. Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.
11. Pregnancy or inability to practice adequate contraception in women of childbearing potential.
12. Evidence of hepatocellular carcinoma: alpha-fetoprotein levels greater than 200 ng/ml and/or liver mass on imaging study that is suggestive of liver cancer.
13. Any other condition, which, in the opinion of the investigators would impede competence or compliance or possibly hinder completion of the study.
14. History of hypersensitivity reactions to metformin.
15. Serum creatinine greater than 1.5 mg/dl in men and greater than 1.4 mg/dl in women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466
- [Derived] Loomba R, Lutchman G, Kleiner DE, Ricks M, Feld JJ, Borg BB, Modi A, Nagabhyru P, Sumner AE, Liang TJ, Hoofnagle JH. Clinical trial: pilot study of metformin for the treatment of non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2009 Jan;29(2):172-82. doi: 10.1111/j.1365-2036.2008.03869.x. Epub 2008 Oct 9. PMID 18945255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 28 adult patients with biopsy-proven NASH were enrolled in the study and 26 completed the 48 weeks of therapy and underwent follow-up metabolic testing, imaging and repeat liver biopsy. 2 patients dropped out were not included in analyses.
Pre-assignment Details: The two drop-outs included a 26-year-old woman who stopped therapy after 12 weeks because she had moved and her employment did not allow time for travel for outpatient visits and a 53-year-old woman who stopped therapy after 24 weeks because of desire to pursue other treatments.
Groups:
- Metformin: Participants will undergo a complete medical examination, a series of lab tests, and a liver biopsy. They will then start taking a single 500-mg tablet of metformin once a day for 2 weeks, then the same dosage twice a day for 2 more weeks, if they tolerate the first dosage. The dosage will increase to 1,000 mg twice a day for the remaining 44 weeks of the study. After 1 year, participants will undergo a repeat medical examination and liver biopsy.
Period: Overall Study
Arm/Group | Metformin
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 17
  Hispanic White | 4
  Asian | 5
  African-American | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Body Mass Index [Number; unit: participants]
  Overweight (BMI=25-30 kg/m^2) | 8
  Obese (BMI=30-40 kg/m^2) | 13
  Severely Obese (BMI greater than 40 kg/m^2) | 5
Glucose tolerance [Number; unit: partcipants] — Impaired glucose tolerance is defined by fasting glucose 110-125 or >=160 mg⁄ dL after 2-h glucose load
  partcipants
    impaired | 8
    not impaired | 18
Diabetes [Number; unit: participants] — Diabetes is defined by a fasting glucose greater or equal to 125 or greater or equal to 200 mg per dL aftera 2-h glucose load.
  participants
    Yes | 7
    No | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in the Histological NASH Activity Index at 48 Weeks Compared With Baseline (Number of Participants in Each Change Category)
Description: Patients under went liver biopsy, metabolic profiling and imaging studies before and at the end 48 weeks of metformin (2000 mg/day) therapy. The primary endpoint is a three point improvement in the histological NASH activity index with a decrease in at least two of the component scores and no worsening of fibrosis or increase in Mallory bodies.
Time Frame: from baseline to 48 Weeks
Measure: Number; unit: participants
Arm/Group | Metformin
Number analyzed (Participants) | 26
participants
  improved (reduced) by greater or equal to 3 points | 9
  improved (reduced) by 1-2 points | 11
  no change | 5
  worsen (increased) | 1
Statistical Analysis 1: Comparison: Metformin; self-controlled comparison of NASH activity index at 48 weeks and baseline. Null hypothesis is "no change"; Test type: Superiority or Other; p < 0.001, paired t-test

2. Secondary Outcome: Change in Serum Alanine Aminotransferase (ALT) Levels From Baseline (Number of Participants in Each Change Category)
Description: Alanine transaminase <42 U/L is considered normal
Time Frame: from baseline to 48 weeks
Measure: Number; unit: participants
Arm/Group | Metformin
Number analyzed (Participants) | 26
participants
  changed to normal from abnormal | 9
  unchanged (normal at beginning) | 4
  unchanged (abnormal at beginning) | 12
  changed to abnormal from normal | 1
Statistical Analysis 1: Comparison: Metformin; self-controlled comparison of serum aminotransferase levels at 48 weeks and baseline. Null hypothesis: No change; Test type: Superiority or Other; p = 0.04, Fisher Exact

3. Secondary Outcome: Change in Insulin Sensitivity (Glucose Tolerance, Homeostatic Model Assessment of Insulin Resistence (HOMA-IR)) From Baseline
Description: HOMA-IR is calculated from Fasting Glucose and Fasting Insulin
Time Frame: from baseline to 48 weeks
Measure: Mean (Standard Deviation); unit: unit
Arm/Group | Metformin
Number analyzed (Participants) | 26
unit | -3.3 (3.2)
Statistical Analysis 1: Comparison: Metformin; Test type: Superiority or Other; p = 0.04, paired t-test

ADVERSE EVENTS:
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 21/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=26)
Weight loss (General disorders) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No